CLINICAL TRIAL: NCT05441722
Title: Feasibility of Neurophysiological Assessments and Exercise Prehabilitation in Breast Cancer Patients Receiving Taxane-based Chemotherapy: a Pilot Randomised Controlled Trial
Brief Title: CIPN in Early Stage Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Gateshead Health NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 262840
Record Dates: First submitted 2022-04-04; First posted 2022-07-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will be invited to perform a bout of supervised moderate-intensity aerobic exercise. Patients receiving chemotherapy with sequential anthracycline-docetaxel will be offered the exercise before each docetaxel-containing infusion, whilst patients receiving weekly paclitaxel will perform the exercise every three weeks during treatment. Each session will comprise of moderate-intensity aerobic exercise on a cycle ergometer. Participants will perform a 5 to 10-minute warm-up.
  Participants will then complete a 30-minute bout at 13-14 RPE whilst. This corresponds to a qualitative description of "somewhat hard" and equates to approximately 60% age-predicted heart rate reserve. Heart rate will be monitored continuously with a Polar heart rate monitor and RPE will be collected every 5-minutes. The resistance on the bike will be reduced if heart rate reserve is > 65% or RPE is > 14 on the 6-20 Borg scale. Each session will finish with a 5 min cool-down at low-intensity (≤ 11 RPE).
  Interventions: Behavioral: Exercise prehabilitation
- Control (No Intervention): Participants allocated to this group will not receive a specific exercise intervention, but will be given a leaflet that provides general physical activity recommendations for cancer patients.
  Recommendations will be based on published guidelines from the American College of Sports Medicine and American Cancer Society.

INTERVENTIONS:
Behavioral: Exercise prehabilitation — Exercise on a cycle ergometer 24 hours before chemotherapy infusion.
  Arms: Exercise

SUMMARY:
Chemotherapy uses anti-cancer drugs to destroy cancer cells and is a common treatment for many cancers. Taxanes are the most widely used chemotherapy drugs given to breast cancer patients. However, taxanes also have toxic side effects. One of the most severe side effects is damage to nerves in the peripheral nervous system; a neurological disorder known as peripheral neuropathy. Common symptoms of peripheral neuropathy are pain, numbness, and tingling in the hands and feet, which can lead to chemotherapy being prematurely discontinued. Unfortunately, treatment options to manage peripheral neuropathy are limited. Exercise has recently been proposed to reduce symptoms, but consistently exercising during chemotherapy is challenging for patients because of treatment-related side effects and fatigue. A more feasible approach may be to exercise on the day before each infusion.

This research includes two linked studies that aim to evaluate whether measuring peripheral nerve function at various timepoints throughout chemotherapy and performing aerobic exercise 24 hours before each infusion is feasible and acceptable to patients. In study 1, the investigators will recruit early stage breast cancer patients, who are scheduled to receive taxanes, from medical oncology outpatient clinics. The investigators will ask consenting participants to make 4 or 5 separate visits to the Hospital at various timepoints throughout chemotherapy, depending on the type of chemotherapy they are prescribed. Each study visit will involve completing some questionnaires as well as tests of peripheral nerve function and functional ability. In phase 2, a new cohort of breast cancer patients undergoing the same chemotherapy regimens will be randomly allocated to an exercise group or a control group. The exercise group will be invited to perform a supervised bout of aerobic exercise (30 min of moderate-intensity on a cycle ergometer) one day before they receive chemotherapy. The findings will lay the foundations for future large-scale research.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed stage IA-IIIC breast cancer.
* Scheduled to receive adjuvant or neoadjuvant chemotherapy with sequential anthracycline-docetaxel or weekly-paclitaxel.
* Willing and able to give written informed consent.
* Understand written and verbal instructions in English.
* American Society of Anaesthesiologists physical status I-III.

Exclusion Criteria:

Pre-existing diabetes mellitus.

* Pregnancy.
* Any sign/symptom of cardiovascular, metabolic or renal disease
* Diagnosed with metastatic breast cancer.
* Previous or existing symptoms of peripheral neuropathy.
* Absolute or relative contraindication to exercise testing and training as defined by the American College of Sports Medicine (ACSM) (38).
* Resting hypertension (≥ 180/100 mmHg) or tachycardia (≥ 100 bpm)
* Pre-existing cardiovascular, musculoskeletal, neurological or psychiatric condition that may affect their ability to complete the testing battery (as determined by the patient's treating Medical Oncologist).
* Internal electrical regulator (cardiac pacemaker or implantable cardioverter defibrillator).
* Previous exposure to taxanes at any time or exposure to other chemotherapy agents known to be associated with neuropathy (e.g., platinum therapy, bortezomib, vinblastine) within one year of starting in the study.
* Currently enrolled in clinical trials involving exercise or pharmacotherapy that could influence CIPN symptoms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | Through study recruitment, predicted time frame of 1 year.
  This is assessed via the number of eligible patients who are invited and give informed consent to participate in the trial.
Reasons for dropout in discontinuing patients | 18 months
  Qualitative- when a participant no longer wants to take part, the reason for drop-out, if given, will be noted.
Retention rates | Up to 18 months
  The number of participants that continue to take part in the study throughout. The retention rates between those who did and did not receive their preferred allocation will then be compared.
Feasibility of measurement procedures | 18 months
  This will be assessed via the number of consented participants who complete baseline and follow-up testing.
Attendance rates (to intervention) | Up to 18 months
  This will be assess by the percentage of exercise interventions that are attended bu participants in the intervention group.
The Physical Activity Enjoyment Scale (PACES) | Up to 18 months
  The Physical Activity Enjoyment Scale is an 18-item scale that assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7- point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it). Eleven items were negatively worded and seven items were positively worded. After reverse scoring the 11 negatively worded items, an overall enjoyment for physical activity score is determined by summing the items, with a range of 18-126 being possible. Higher scores indicate higher enjoyment.
Adverse events | Up to 18 months
  The number and type of adverse events experienced by participants will be noted to assess safety, along with exploring reasons for discontinuing exercise.

SECONDARY OUTCOMES:
European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy twenty-item scale (QLQ-CIPN20) | Up to 18 months
  The QLQ-CIPN20 contains 20 items assessing sensory (9 items), motor (8 items), and autonomic symptoms (3 items). Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), individuals indicate the degree to which they have experienced sensory, motor, and autonomic symptoms during the past week. Sensory raw scale scores range from 1 to 36, motor raw scale scores range from 1 to 32, and autonomic raw scale scores range from 1 to 12 for men and 1-8 for women (erectile function item is excluded). All scale scores are linearly converted to a 0-100 scale, with higher scores indicating more symptom burden.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Up to 18 months
  The FACIT-Fatigue scale is a 13-item questionnaire originally designed to assess fatigue/tiredness and its impact on daily functioning in people with cancer; it has now been evaluated in other chronic diseases. Each item's response option uses a 5-point scale ranging from "not at all" to "very much." The total FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue.
Pain Quality Assessment Scale (PQAS). | Up to 18 months
  Participants are asked to rate the severity of each of the 20 pain domains using 0 to 10 numerical rating scales, where 0="no pain" or "not (sensation/item)" and 10="the most (descriptor) pain sensation imaginable."
Godin Leisure-Time Exercise Questionnaire. | Up to 18 months
  The GLTEQ measures the frequency of strenuous, moderate, and mild LTPA performed for periods of 15 min or more over a usual week.
Functional Assessment of Cancer Therapy-Breast (FACT-B) | Up to 18 months
  The FACT-B is a breast cancer-specific HRQoL instrument of the FACIT system. The 37-item English and (simplified) Chinese FACT-B version 4 are divided into five subscales, namely physical (PWB), social/family (SWB), emotional (EWB), functional well-beings (FWB), and the additional concerns for breast cancer (BCS). Each item is rated on a 5-point Likert scale. Negatively worded items were recoded such that a higher score indicates a better HRQoL. The FACT-B total score is the sum of scores of all five subscales.
Physician-reported CIPN | Up to 18 months
  Graded by the treating Medical Oncologist using the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) grading scale. CIPN is rated from 1 to 5 depending on the severity.
Body mass | Up to 18 months
  Body mass will be measured to the nearest 0.1 kg using a calibrated digital scale.
Waist circumference | Up to 18 months
  Waist circumferences will be measured to the nearest 0.1 cm using a nonstretching measuring tape.
Height | Up to 18 months
  Standing height will be measured to the nearest 0.1 cm with a free-standing stadiometer
Hip circumference | Up to 18 months
  Hip circumferences will be measured to the nearest 0.1 cm using a nonstretching measuring tape.
Short Physical Performance Battery (SPPB) | Up to 18 months
  The SPPB is a composite measure of standing balance, gait speed and chair sit-to-stand tests. The tests include: 1) the ability to stand for up to 10 seconds with feet positioned side-by-side, semi-tandem and tandem, 2) time to complete a 4-m walk at usual pace, and 3) number of sit-to-stands achieved in 30 s.
Tandem walk test | Up to 18 months
  Participants walk for 10 steps, heel-to-toe, without spaces between the steps. Two trials will be performed, one with eyes open and one with eyes closed. The maximum number of consecutive steps will be recorded (maximum of 10). Errors will include taking a side step, making a space between the feet, and opening the eyes during the eyes closed trial.
Maximal isometric grip strength | Up to 18 months
  Participants will squeeze an analogue hand grip dynamometer (Takei Scientific Instruments Ltd., TKK 183 5001 Grip-A, Tokyo, Japan) as hard as possible for 2-3 s. Three maximal trials will be performed on each hand, with the highest score used for analysis.
Vibration perception (128 Hz tuning fork) | Up to 18 months
  The "on-off" method will be used. The tuning fork is struck before being applied to the bony prominence situated at the dorsum of the hallux in the feet, and pollux in the hand, both just proximal to the nail bed. The patient is asked to indicate whether they feel a vibration. The patient is then asked to indicate when the vibration has stopped. One point is assigned for each vibration sensation perceived, and another point is assigned if the correct timing of the dampening of the vibration is perceived. This procedure is repeated twice on each foot and each hand. The overall score ranges from 0 to 8.
Touch perception (Semmes-Weinstein 10g Monofilament) | Up to 18 months
  The monofilament is lightly pressed against the skin for three seconds so that it buckles into a C shape. The patient is asked to indicate whether they feel the touch. Four sites will be tested on each foot: the plantar surface of the hallux, the plantar surfaces of the first, third and fifth metatarsal heads. This will also be conducted in equivalent locations in the hand. One point is assigned for each senate site, hence, the overall score ranges from 0 to 8 for each of hands and feet.
Temperature perception (Tip Therm GmbH, Brueggen, Germany) | Up to 18 months
  The Tip-therm is a pen-like device with a metal cylinder on one end and a polymer cylinder on the other end. The metal side feels colder than the polymer side due to the thermal conductivity property of the material. Both ends of the device are applied to the dorsal surface of the foot between the base of the hallux and the second toe and at the dorsum of the second metacarpal in the hand between the ring and index fingers, for three seconds. The patient is asked which surface they felt was colder. One point is assigned if the correct temperature is perceived. This procedure is repeated twice on each foot and each hand, with an overall score assigned to each patient that ranges from 0 to 4 for each of hands and feet.
Peripheral Nerve Function | Up to 18 months
  H-reflex and M-wave elicited in the soleus muscle. An H-reflex and M-wave recruitment curve will be plotted and changes in Hmax/Mmax and H reflex latency will be extracted.
Sway- accelerometer | Up to 18 months
  Participants will complete the test wearing a wireless tri-axial accelerometer (Delsys, Inc). The accelerometer will be located at the level or the posterior superior iliac spine. The pen will be at the same height and record the displacement of the body by tracing a line on a sheet of paper. Participants will be asked to stand barefoot 'as still as possible without talking' for 30 seconds. This will be conducted while the patient is standing on both legs. Standing balance will be quantified as postural sway path length.
Sway - swaymeter | Up to 18 months
  The swaymeter involves wearing a belt that will have an inflexible rod attached and a vertically mounted pen at the end of the rod. The rod will be located at the level or the posterior superior iliac spine. The pen will be at the same height and record the displacement of the body by tracing a line on a sheet of paper. Participants will be asked to stand barefoot 'as still as possible without talking' for 30 seconds. This will be conducted while the patient is standing on both legs. Standing balance will be quantified as postural sway path length.
Habitual physical activity | Up to 18 months
  Step counts will be noted via a pedometer and participants will be asked to keep an exercise diary.
Interviews of participants | Up to 18 months
  Questions will relate to acceptability of the intervention, including barriers experienced that impacted their ability to complete the intervention, their attitudes towards exercising during chemotherapy treatment and how well they were able to integrate the exercise sessions into day/life.
9-Hole Peg Test | Up to 18 months
  Participants will be provided with a 9-Hole Peg Test kit, consisting of 9 6mm x 30mm wooden dowels and three lines of three holes (9 in total). The participants will be asked to place the wooden dowels into the holes in any order until all the holes are filled, and then immediately remove them one at a time, returning them to the container provided. This test will be done using twice using their dominant hand and twice using the non-dominant hand. For familiarisation, an additional two tests per hand will be performed in the first assessment visit.

CONTACTS AND LOCATIONS:
Overall Officials: John Temesi, PhD, Principal Investigator — Northumbria University
Locations (1):
- Queen Elizabeth Hospital, Gateshead, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The research team supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov. Upon reporting and publication of tall study outcomes deidentified individual participant data will be released to investigators. Requests may be made to: rosiered.brownson-smith@northumbria.ac.uk.
Supporting Information: Study Protocol, SAP, ICF